CLINICAL TRIAL: NCT02270151
Title: Improving DEtection of Atrial fibriLlation in Primary Care With the MyDiagnostick
Acronym: IDEAL-MD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Monika Hollander, MD, PhD, Monika Hollander, MD, PhD, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 14-163/C
Record Dates: First submitted 2014-09-04; First posted 2014-10-21 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Screening; Primary care; Diagnostic
MeSH Terms: conditions — Atrial Fibrillation; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MyDiagnostick (Active Comparator): Everyone aged 65 years or over, who visits the GP practice will be screened for AF with the MyDiagnostick. When the device indicates a positive result, the single lead ECG will be assessed to confirm/reject the diagnosis. Every new case of diagnosed AF will be evaluated for further treatment by the general practitioner.
  Interventions: Device: MyDiagnostick
- Control (No Intervention): Control arm will perform care as usual with selective screening by feeling the pulse.

INTERVENTIONS:
Device: MyDiagnostick — Diagnostick strategy with MyDiagnostick
  Arms: MyDiagnostick

SUMMARY:
Atrial fibrillation (AF) is the most common arrhythmia and a common cause of stroke. AF can be asymptomatic and remain undiagnosed. Both the prevalence of AF and the proportion of strokes related to undetected AF increases with ageing. If AF is timely diagnosed and treated accordingly with anticoagulants, disabling strokes can be prevented. In order to help physicians in diagnosing atrial fibrillation, the MyDiagnostick was developed. It is a CE certified device that is safe, user friendly and easy to use. This device is capable of detecting or excluding AF within one minute by providing a registration of lead I of the ECG.

The investigators aim to perform a 2-arm cluster randomized diagnostic trial among patients aged 65 years and over who visit the general practice. In total the investigators will include 42 general practices of which they randomly assign 21 to the MyDiagnostick arm and 21 to the control arm. All persons aged 65 years and over who visit the general practice in the MyDiagnostick arm will be asked to hold the device every time they visit the surgery during one year.

The number of newly detected cases of AF with the diagnostic screening strategy with MyDiagnostick (MyDiagnostick arm) will be compared to care as usual (control arm). Also, the number of patients treated with anticoagulants according CHA2DS2-VASc score will be compared between both arms. Finally, the investigators will assess the number of major adverse cardiovascular events (MACE), intracerebral hemorrhages and other major hemorrhages, and all-cause mortality between the arms. End points will be assessed blinded to allocation.

The investigators hypothesise that the MyDiagnostick improves the diagnosis of atrial fibrillation in primary care and with accordingly treatment will reduce adverse outcomes.

DETAILED DESCRIPTION:
In a recent validation study performed in 200 patients visiting a cardiology outpatient clinic, the sensitivity was 100%, and specificity 96.4% with the MyDiagnostics as compared to a 12-lead ECG. Adequate comparison of this device with accordingly treatment with care as usual is needed before large scale implementation in the primary care setting can be advocated.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling persons visit the GP and aged 65 years of over

Exclusion Criteria:

* Terminal illness of such severity that anticoagulation is considered to be not appropriate in case of newly detected atrial fibrillation
* Acute situation in which GP should act instantly
* Patients with a history of AF

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 16000 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Newly detected cases of AF | One year
  For our primary outcome the investigators will calculate the number of atrial fibrillation as detected with MyDiagnostick (MyDiagnostick arm) as compared to care as usual in primary care (control arm)

SECONDARY OUTCOMES:
Adequate treatment of AF according the CHA2DS2-VASc score | one year
  The investigators will compare anticoagulant treatment in newly detected AF patients in the MyDiagnostick with the number of those receiving anticoagulant treatment in new AF cases in the control arm
Major cardiovascular events and all cause mortality | one year
  The investigators will compare major cardiovascular events (ischemic strokes, intracerebral hemorrhages and other major hemorrhages, myocardial infarction, CABG, PCA), and all cause mortality between the MyDiagnostick arm and the control arm within one year after the start of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Frans H Rutten, MD PhD, Principal Investigator — Julius Center, UMC Utrecht; Arno W Hoes, MD PhD prof, Study Chair — Julius Center, UMC Utrecht; Monika Hollander, MD PhD, Principal Investigator — Julius Center, UMC Utrecht
Locations (1):
- GP practices, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Result] Go AS, Hylek EM, Phillips KA, Chang Y, Henault LE, Selby JV, Singer DE. Prevalence of diagnosed atrial fibrillation in adults: national implications for rhythm management and stroke prevention: the AnTicoagulation and Risk Factors in Atrial Fibrillation (ATRIA) Study. JAMA. 2001 May 9;285(18):2370-5. doi: 10.1001/jama.285.18.2370. PMID 11343485
- [Result] Heeringa J, van der Kuip DA, Hofman A, Kors JA, van Herpen G, Stricker BH, Stijnen T, Lip GY, Witteman JC. Prevalence, incidence and lifetime risk of atrial fibrillation: the Rotterdam study. Eur Heart J. 2006 Apr;27(8):949-53. doi: 10.1093/eurheartj/ehi825. Epub 2006 Mar 9. PMID 16527828
- [Result] Jorgensen HS, Nakayama H, Reith J, Raaschou HO, Olsen TS. Acute stroke with atrial fibrillation. The Copenhagen Stroke Study. Stroke. 1996 Oct;27(10):1765-9. doi: 10.1161/01.str.27.10.1765. PMID 8841326
- [Result] Hart RG, Pearce LA, Aguilar MI. Meta-analysis: antithrombotic therapy to prevent stroke in patients who have nonvalvular atrial fibrillation. Ann Intern Med. 2007 Jun 19;146(12):857-67. doi: 10.7326/0003-4819-146-12-200706190-00007. PMID 17577005